CLINICAL TRIAL: NCT05356039
Title: Survival, Quality of Life and Resectability in Locally Advanced Pancreatic Cancer - a Multicenter Prospective Observational Study
Brief Title: Survival, Quality of Life and Resectability in Locally Advanced Pancreatic Cancer
Acronym: SQUARE
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: University Hospital, Linkoeping (Other); Lund University Hospital (Other); Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); University Hospital, Umeå (Other)
Responsible Party: Sponsor
Other Study IDs: UmU-square
Record Dates: First submitted 2022-03-28; First posted 2022-05-02 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Pancreas Cancer; Pancreas Neoplasm; Pancreas Disease; Pancreas Adenocarcinoma; Surgery; Chemotherapy Effect; Quality of Life; Locally Advanced Pancreatic Adenocarcinoma; Borderline Resectable Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma biobanking. Tissue Microarray Construction from formalin fixed paraffin embedded tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess overall survival, quality of life and resection rates in locally advanced pancreatic cancer

DETAILED DESCRIPTION:
This is a multicenter pragmatic prospective observational study including Nordic hospitals treating patients with borderline resectable and locally advanced pancreatic cancer. Eligibility will be assessed at regional multidisciplinary tumor boards. Patients with borderline resectable and locally advanced (non-endocrine) pancreatic cancer according to the National Comprehensive Cancer Network (NCCN) and the International Study Group of Pancreatic Surgery (ISGPS) are eligible for inclusion. The study is observational. Quality of life will be assessed in all study participants. The primary outcomes are exploration rates, resection rates and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected invasive pancreatic primary tumor
* Tumor classified as borderline resectable or locally advanced disease according to NCCN guidelines

Exclusion Criteria:

* Suspected endocrine tumor
* Suspected non-pancreatic periampullary tumor
* Distant metastasis
* Age < 18 years
* Patient unable to understand verbal or written information interfering with informed consent or treatment
* Mental or organic disorder interfering with informed consent or treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed or suspected non-endocrine invasive pancreatic primary tumor that is classified as borderline resectable or locally advanced disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Median Overall Survival | From date of inclusion until the date of death from any cause, assessed up to 72 months
  Median overall survival for patients with locally advanced pancreatic cancer stratified for treatment allocation
Resection | From the time of inclusion to end of study follow up or date of death from any cause, whichever came first, up to 72 months
  Rates of resection among patients with locally advanced pancreatic cancer stratified for treatment allocation

SECONDARY OUTCOMES:
Oncological treatment compliance | From the time of inclusion to end of study follow up or date of death from any cause, whichever came first, up to 72 months
  Number of patients that complete a started oncological treatment and are able to complete regimen
Chemotherapy response | From the time of inclusion to end of study follow up or date of death from any cause, whichever came first, up to 72 months
  Percentage within each RECIST strata
Predictors of resectability | From the time of inclusion to end of study follow up or date of death from any cause, whichever came first, up to 72 months
  Logistic regression models assessing predictors of resectability
Quality of Life at baseline | At first visit/inclusion
  Quality of life assessed with EORTC QLQ C30 focused on self-reported Global Health Score ranging from 1 to 7 where a higher number indicates better self-experienced health
Quality of Life at 3 months after inclusion | Quality of Life at 3 months after inclusion
  Quality of life assessed with EORTC QLQ C30 focused on self-reported Global Health Score ranging from 1 to 7 where a higher number indicates better self-experienced health
Quality of Life at 6 months after inclusion | Quality of Life at 6 months after inclusion
  Quality of life assessed with EORTC QLQ C30 focused on self-reported Global Health Score ranging from 1 to 7 where a higher number indicates better self-experienced health
Quality of Life at 9 months after inclusion | Quality of Life at 9 months after inclusion
  Quality of life assessed with EORTC QLQ C30 focused on self-reported Global Health Score ranging from 1 to 7 where a higher number indicates better self-experienced health
Quality of Life at 12 months after inclusion | Quality of Life at 12 months after inclusion
  Quality of life assessed with EORTC QLQ C30 focused on self-reported Global Health Score ranging from 1 to 7 where a higher number indicates better self-experienced health
Quality of Life at 24 months after inclusion | Quality of Life at 24 months after inclusion
  Quality of life assessed with EORTC QLQ C30 focused on self-reported Global Health Score ranging from 1 to 7 where a higher number indicates better self-experienced health

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Clinic at Umeå University Hospital, Umeå, Sweden